CLINICAL TRIAL: NCT06516367
Title: Development and Validation of a New Tool for Simultaneous Screening of Malnutrition, Sarcopenia, and Cachexia in Older Adults
Brief Title: Screening Tool for Malnutrition, Sarcopenia, and Cachexia
Acronym: ASUST-MSC
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doha Rasheedy, Professor of Geriatrics and Gerontology, Ain Shams University
Other Study IDs: Ain Shams Screening tools
Record Dates: First submitted 2024-07-03; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Malnutrition; Sarcopenia; Cachexia
Keywords: screening; older adult; malnutrition; cachexia; sarcopenia
MeSH Terms: conditions — Malnutrition; Sarcopenia; Cachexia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ain Shams University Screening Tool for Malnutrition, Sarcopenia, and Cachexia (ASUST-MSC) — 25 items dichotomous questionnaire
  Other Names: bioelectrical impedence analysis; handheld dynamometer

SUMMARY:
There is an accumulating evidence of the overlap and frequent co-occurrence of twasting conditions in older adults. Those conditions include malnutrition, sarcopenia, and cachexia, Therefore , a tool capable of simultaneously screening for all three conditions is imperative. In this study, we developed and validated a new tool for the simultaneous screening of muscle wasting diseases in older adults. The diagnostic accuracy of the new tool was compared to other validated screening tools including the Mini Nutritional Assessment-Short Form (MNA-SF), the Short Nutritional Assessment Questionnaire (SNAQ), and the Simple Questionnaire to Rapidly Diagnose Sarcopenia (SARC-F).

ELIGIBILITY:
Inclusion Criteria:

* Participants Aged 65 years and older, who agree to participate

Exclusion Criteria:

* Patients with critical illness.
* Patients with severe cognitive, hearing or visual impairment hindering proper communication
* Patients with physical disability that interfere with physical performance assessment or hand grip measurement
* Patient with any contraindication of to the use of BIA) e.g. presence of a pacemaker, other implanted electrical devices, or metal implants, volume overload

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: 300 older participants aged 60 years old and above who were admitted to Ain Shams University Hospitals or interviewed at the hospital clinic
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
reliability of a new tool for the simultaneous screening of muscle wasting diseases in older adults | 10 months
  Relaibility; Cronbach's alpha coefficient was used to evaluate the internal consistency.
validity of a new tool for the simultaneous screening of muscle wasting diseases in older adults | 10 months
  Validity; Spearman's correlation coefficient was used to examine construct validity of the new tool

SECONDARY OUTCOMES:
The diagnostic accuracy of the new tool | 10 months
  The Receiver operating curve was plotted to detect the area under curve of the new tool, for diagnosing muscle wasting diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No